CLINICAL TRIAL: NCT06078124
Title: Sibling-Support for Adolescent Girls (SSAGE): A Whole-family, Gender Transformative Approach to Preventing Mental Illness Among Forcibly Displaced Adolescent Girls
Brief Title: Sibling-Support for Adolescent Girls (SSAGE)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Universidad de Los Andes (Unknown); Women's Refugee Commission (Unknown); National Institutes of Health (NIH) (NIH); Mercy Corps (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R34MH134078-01 (NIH)
Record Dates: First submitted 2023-09-28; First posted 2023-10-11 (Actual); Results first posted 2025-07-20 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Anxiety; Depression; Mental Illness
Keywords: Mental illness; Adolescent girls; Forcibly displaced populations; Randomized-controlled trial; Implementation science; Family functioning; Gender inequity
MeSH Terms: conditions — Anxiety Disorders; Depression; Mental Disorders | interventions — Emergency Service, Hospital

STUDY DESIGN:
Intervention Model Description: A hybrid type 1 effectiveness-implementation pilot randomized-controlled trial with one treatment arm and one control arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sibling Support for Adolescent Girls in Emergencies (SSAGE) (Experimental): Participants in this arm will participate in the Sibling Support for Adolescent Girls in Emergencies (SSAGE) intervention, along with three family members, for twelve weeks
  Interventions: Behavioral: Sibling Support for Adolescent Girls in Emergencies
- Control arm (No Intervention): Care as usual

INTERVENTIONS:
Behavioral: Sibling Support for Adolescent Girls in Emergencies — The Sibling Support for Adolescent Girls in Emergencies (SSAGE) intervention is a gender-transformative, 12-week program utilizing a "whole family approach" wherein an adolescent girl, her male sibling, and a male and female caregiver participate in sessions that are age- and gender-specific and combined with family-wide discussions of session learnings. The sessions are interactive, engaging, and promote self-reflection and discussion on topics such as power, gender, interpersonal communication, and healthy relationships. Given the whole-family approach, SSAGE addresses intersections between spousal relationships, caregiver-child relationships, and relationships between siblings, as they pertain to supporting the mental health and psychosocial well-being of adolescent girls.
  Other Names: SSAGE
  Arms: Sibling Support for Adolescent Girls in Emergencies (SSAGE)

SUMMARY:
Forcibly displaced adolescents face increased risks for mental illness and distress, with adolescent girls disproportionately affected in part due to the heightened gender inequity that often accompanies forced displacement. Although the family unit has the potential to prevent mental illness and promote healthy development in adolescents, few family interventions have employed a gender transformative approach or included male siblings in an effort to maximize benefits for adolescent girls. Therefore, the investigators propose to assess an innovative whole-family and gender transformative intervention-Sibling Support for Adolescent Girls in Emergencies (SSAGE)-to prevent mental health disorders among adolescent girls in Colombia who were recently and forcibly displaced from Venezuela. The proposed R34 study will adapt the SSAGE curriculum through human-centered design with a range of stakeholders, including Venezuelan refugees, Colombian returnees and relevant civil society organizations. The proposed study will then employ a hybrid type 1 effectiveness-implementation pilot randomized control trial (RCT) to test the program's effectiveness and mechanistic pathways as well as to explore determinants of implementation in order to establish the feasibility, acceptability, and fidelity of SSAGE. To address these aims, the investigators will enroll 180 recently arrived, forcibly displaced adolescent girls in an RCT and examine the program's effectiveness on the prevention of mental illness (through reduction in anxiety, depression, interpersonal sensitivity, and somatization symptoms) one-month post-intervention. The investigators will use contextually adapted and piloted measures to collect additional data on the hypothesized mechanistic pathways, including family attachment, gender equitable family functioning, self-esteem, and coping strategies. The implementation evaluation will employ mixed methods to assess the program's feasibility, acceptability, fidelity and barriers and facilitators to successful implementation. Potential findings can support humanitarian program implementation, as well as inform policy to support adolescent girls' mental health and to prevent the myriad disorders that can arise as a result of exposure to displacement, conflict, and inequitable gender norms in their households and communities.

ELIGIBILITY:
Inclusion Criteria:

* Live with a male and female caregiver and an adolescent male sibling or relative
* Immigrated to Colombia within the last year
* Are available, along with their family members, to participate in the SSAGE intervention for three months
* Are available to participate in survey questionnaires immediately before and one month after the intervention

Exclusion Criteria:

* None

Ages: 13 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 186 (Actual)
Dates: Start 2024-08-05 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Stark, DrPH, Principal Investigator — Washington University School of Medicine
Locations (1):
- Los Andes University, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: Yes
De-identified questionnaire data will be shared beginning 3 months and ending 5 years following article publication with qualified researchers who have a research question appropriate to the data and of potential benefit to forcibly displaced adolescent girls. Deidentified data will only be provided in aggregate after completion of a data use agreement. Requests should be directed to lindsaystark@wustl.edu. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Qualified researchers who have a research question appropriate to the data and of potential benefit to forcibly displaced adolescent girls will be granted access to the data. Requests should be directed to lindsaystark@wustl.edu. Deidentified data will only be provided in aggregate after completion of a data use agreement.

RESULTS

PARTICIPANT FLOW:
Groups:
- Sibling Support for Adolescent Girls in Emergencies (SSAGE): Participants in this arm will participate in the Sibling Support for Adolescent Girls in Emergencies (SSAGE) intervention, along with three family members, for twelve weeks.
  Sibling Support for Adolescent Girls in Emergencies: The Sibling Support for Adolescent Girls in Emergencies (SSAGE) intervention is a gender-transformative, 12-week program utilizing a "whole family approach" wherein an adolescent girl, her male sibling, and a male and female caregiver participate in sessions that are age- and gender-specific and combined with family-wide discussions of session learnings. The sessions are interactive, engaging, and promote self-reflection and discussion on topics such as power, gender, interpersonal communication, and healthy relationships. Given the whole-family approach, SSAGE addresses intersections between spousal relationships, caregiver-child relationships, and relationships between siblings, as they pertain to supporting the mental health and psychosocial well-being of adolescent girls.
  Although multiple family members may participate in the program, the study only enrolls adolescent girls. Family members are not part of the study and data are only collected from adolescent girls.
Period: Overall Study
Arm/Group | Sibling Support for Adolescent Girls in Emergencies (SSAGE) | Control Arm
Started | 93 | 93
Completed | 79 | 79
Not Completed | 14 | 14
Not completed — Lost to Follow-up | 14 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sibling Support for Adolescent Girls in Emergencies (SSAGE) | Control Arm | Total
Number analyzed (Participants) | 93 | 93 | 186
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.84 (1.96) | 15.82 (1.79) | 15.83 (1.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 93 | 186
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 93 | 93 | 186
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 93 | 93 | 186
Region of Enrollment [Count of Participants; unit: Participants]
  Colombia | 93 | 93 | 186
Nationality [Count of Participants; unit: Participants]
  Colombian | 9 | 7 | 16
  Venezuelan | 84 | 86 | 170
Currently in school [Count of Participants; unit: Participants] | 77 | 76 | 153

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 Level 1 Cross-Cutting Symptom
Description: This measure initially includes 25 items and assesses the presence and severity of several psychiatric symptom domains in children and adolescents over the last two weeks. 19 of the items are rated on a 5-point scale (0=none/never; 1=slight/rare; 2=mild/several days; 3=moderate/more than half the days; and 4=severe/almost daily). Questions on suicide ideation, suicide attempts, and substance use are rated on a 2-point scale of yes/no. The included symptoms represent 12 domains of mental disorders: somatic symptoms, sleep problems, inattention, depression, anger/irritability (measured together), mania, anxiety, psychosis, repetitive thoughts and behaviors, substance use, and suicide ideation/attempts. Generally, a respondent is flagged as requiring further inquiry for a given domain if they answered '2' or higher on at least one of the symptoms in each respective domain. As such, this outcome is operationalized as 12 dichotomous variables reflecting the 12 domains.
Time Frame: Up to 2 weeks following the end of the 12 week intervention
Population: Outcomes for the 158 adolescent girls measured at endline. All girls are 13-19 years old and are forcibly displaced.
Measure: Count of Participants; unit: Participants
Arm/Group | Sibling Support for Adolescent Girls in Emergencies (SSAGE) | Control Arm
Number analyzed (Participants) | 79 | 79
Participants
  Somatic symptoms | 44 | 42
  Sleep problems | 24 | 28
  Inattention | 50 | 41
  Depression | 39 | 43
  Anger/irritability | 38 | 40
  Mania | 31 | 22
  Anxiety | 38 | 40
  Psychosis | 22 | 18
  repetitive thoughts and behaviors | 57 | 47
  Substance use | 21 | 17
  Suicide ideation/attempts | 31 | 30

2. Primary Outcome: Revised Children's Anxiety and Depression Scale (RCADS)-25
Description: This scale assesses symptoms of depression and anxiety over the past two weeks in children and adolescents using 25 items. Items are scored on a 4-point scale (0-never; 1-sometimes; 2-often; and 3-always) for the last two weeks. The sum of all item scores are then converted into t-scores based on gender and age. Ranges are as follows: t-score<65 is normal range; >=65 and <=69 is borderline clinical; and >=70 is clinical range.
Time Frame: Up to 2 weeks following the end of the 12 week intervention
Population: Participants are forcibly displaced adolescent girls ages 13-19 years old. Measures were taken at endline (post-intervention) for 79 treatment and 79 control participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Sibling Support for Adolescent Girls in Emergencies (SSAGE) | Control Arm
Number analyzed (Participants) | 79 | 79
Participants
  Normal range | 58 | 61
  Borderline clinical | 6 | 4
  Clinical range | 15 | 14

3. Secondary Outcome: Family Attachment and Changeability Index (FACI-8) (Modified)
Description: We employed a modified version of the FACI8. The FACI8 is traditionally a 16-item scale where each item is scored using a 4-point Likert scale of how frequently the event occurs in the last 2 weeks (1-Never; 2-Sometimes; 3-Most of the time; 4-Always). During baseline training, it was determined that four of the items in the traditional FACI8 were not reliable or valid in our study setting. As such, a 12-item version was employed. The modified FACI8 consists of two subscales: Attachment and Changeability. The attachment subscale includes 7 items and the changeability subscale comprises 5 items. Subscale scores are created by summing the relevant item responses. Unfortunately, there was a tech issue with one of the changeability items at endline and data were not collected for that item. As such, we removed that item from the changeability subscale to preserve comparability with baseline. The final score for attachment can be 7-28 and changeability from 4-16. Higher scores are better.
Time Frame: Up to 2 weeks following the end of the 12 week intervention
Population: Note to ClinicalTrials.gov: Unfortunately, this scale was not found to be valid or reliable with our study population and we therefore did conduct any analysis with this measure. As such, we do not feel it is appropriate for others to derive any conclusions from the results for these measures.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sibling Support for Adolescent Girls in Emergencies (SSAGE) | Control Arm
Number analyzed (Participants) | 79 | 79
units on a scale
  Attachment subscale | 20.23 (3.17) | 20.67 (2.94)
  Changeability subscale | 11.18 (2.74) | 11.16 (2.66)

4. Secondary Outcome: Rosenberg Self-Esteem Scale
Description: The Rosenberg Self-Esteem Scale is a 10-item scale that measures positive and negative feelings about the self to create a measure of overall self-worth. Items are scored using a 4-point Likert scale signaling level of agreement with each statement, from strongly agree to strongly disagree. Five items are reverse coded. The final score can take a value from 10 to 40, with higher scores indicating greater self-esteem. The scale asks about the last two weeks and the measure was taken up to 2 weeks following the end of the 12 week intervention.
Time Frame: Up to 2 weeks following the end of the 12 week intervention
Population: 158 adolescent girls who participated in a pilot-RCT of SSAGE. Participants are 13-19 years old and are forcibly displaced within Colombia.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sibling Support for Adolescent Girls in Emergencies (SSAGE) | Control Arm
Number analyzed (Participants) | 79 | 79
units on a scale | 30.09 (3.16) | 29.87 (3.16)

5. Secondary Outcome: Kidcope
Description: Kidcope is a 15-item checklist designed to measure cognitive and behavioural coping in children and adolescents. It measures the frequency of 15 coping strategies, including: problem-solving, distraction, social support, social withdrawal, cognitive restructuring, self-criticism, blaming others, emotional expression, wishful thinking and resignation. Items rare scored on a 4-point scale (0 = "Not at all" to 3 = "Almost all the time"). The final measure is operationalized as 15 dichotomous indicators, where a '1' signals the participant used that coping strategy at least sometimes in the last two weeks for a stressor and a '0' means the participant never used the coping mechanism in the last two weeks.
Time Frame: A stressor that occurred in the last two weeks; measurement taken up to 2 weeks following the end of the 12 week intervention
Population: 13-19 year-old girls, half of whom participated in the SSAGE intervention. All participants are forcibly displaced.
Measure: Count of Participants; unit: Participants
Arm/Group | Sibling Support for Adolescent Girls in Emergencies (SSAGE) | Control Arm
Number analyzed (Participants) | 79 | 79
Participants
  Thought about som ething else or tried to forget | 67 | 64
  Did something to distract self like watch TV or play a game | 67 | 72
  Stayed away from people and kept feelings to self | 57 | 66
  Handled the situation on own | 66 | 65
  Tried to see bright side of things and/or focus on something good | 72 | 75
  Blamed self for causing problem | 36 | 39
  Blamed someone else for putting through problem | 27 | 23
  Thought of ways to solve problem | 75 | 71
  Tried to solve problem on own | 67 | 69
  Screamed, cried, or hit something | 37 | 40
  Tried to calm down byt talking to self, praying, taking a walk | 70 | 73
  Kept thinking and wishing stressor never happened | 57 | 54
  Kept wishing could change what had happened | 60 | 59
  Turned to family, friends, or other adults to help feel better | 60 | 56
  Just accepted the problem because knew there was nothing to do about it | 64 | 60

ADVERSE EVENTS:
Time Frame: ~12-14 weeks following enrollment/baseline data collection, which also when endline data collection took place.
Arm/Group | Sibling Support for Adolescent Girls in Emergencies (SSAGE) | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/93 | 0/93
Serious Adverse Events (participants affected / at risk) | 0/93 | 0/93
Other Adverse Events (participants affected / at risk) | 0/93 | 0/93

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2024-07-12): https://cdn.clinicaltrials.gov/large-docs/24/NCT06078124/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-20): https://cdn.clinicaltrials.gov/large-docs/24/NCT06078124/SAP_001.pdf
  • Informed Consent Form (2024-07-15): https://cdn.clinicaltrials.gov/large-docs/24/NCT06078124/ICF_002.pdf